CLINICAL TRIAL: NCT03196934
Title: A Multicenter, Open-label, Flexible Dose Study to Assess the Long-term Safety of Pharmaceutical Cannabidiol Oral Solution as an Adjunctive Treatment for Pediatric Subjects With a Treatment-resistant Seizure Disorder Who Complete INS011-14-029 or Part A of INS011-15-054
Brief Title: Expanded Use of Cannabidiol Oral Solution
Status: No longer available | Type: Expanded Access
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MulticareHSRI
Record Dates: First submitted 2017-03-21; First posted 2017-06-23 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Cannabidiol oral solution — Cannabidiol; Pharmacological class of drug

SUMMARY:
To allow subjects who have completed Insys 030 extension study to continue to take Cannabidiol oral solution.

DETAILED DESCRIPTION:
To allow subjects who have completed Insys 030 extension study (A multicenter, open-label, flexible dose study to assess the long-term safety of pharmaceutical Cannabidiol Oral Solution as an adjunctive treatment for pediatric subjects with a treatment-resistant seizure disorder who complete INS011-14-029 or Part A of INS011-15-054) to continue to take Cannabidiol oral solution.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the Insys 030 protocol
2. Compliant in drug study procedures
3. Non-pregnant females of child bearing age, willing to utilize a double-barrier method of birth control during treatment and for 30 days after treatment has ended

Exclusion Criteria:

1. Failure to follow study procedures in Insys 030
2. Pregnant females

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult